CLINICAL TRIAL: NCT01521247
Title: Implementation of a Pediatric-to-adult Asthma Transition Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Warren Davidson, Principal Investigator, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: AJMG-2010
Record Dates: First submitted 2012-01-23; First posted 2012-01-30 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Asthma; Education
Keywords: Asthma; Transition program; Pediatric; Adult
MeSH Terms: conditions — Asthma | interventions — Referral and Consultation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): Usual care.
- Asthma Transition Program (Other): Asthma Transition Program
  Interventions: Other: Asthma Transition Program

INTERVENTIONS:
Other: Asthma Transition Program — Asthma Education.
  Other Names: Asthma Education and Referral.
  Arms: Asthma Transition Program

SUMMARY:
Despite the clear and often stated need, a formal transition program does not exist for asthma patients as they move from pediatric to adult care in Western Canada. This population is not having their health care needs met. The investigators proposed study would evaluate a well structured transition program designed to facilitate continuity of care for this at risk patient population.

Primary hypothesis: A pediatric-to-adult asthma transition program will improve the asthma-specific quality of life of young asthma patients in the Calgary area over a 1 year period.

Secondary hypothesis: A pediatric-to-adult asthma transition program will improve asthma control, decrease asthma exacerbations, and reduce health care utilization in young asthma patients in the Calgary area over a 1 year period.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of asthma (as confirmed by a pediatric respirologist or pediatrician with asthma expertise, and including evidence of variable airflow obstruction, bronchial hyperresponsiveness, airway inflammation, and/or response to therapy)

Exclusion Criteria:

* patients who are known to be non-adherent within the Calgary Regional Pediatric Asthma Clinic (defined as >50% missed appointments over a 2 year period)
* patients unable to complete pulmonary function testing
* patients with a history of significant respiratory comorbid conditions (including history of cystic fibrosis, alpha-1 antitrypsin deficiency, and lung transplant - rhinosinusitis patients will not be excluded)
* patients unable to provide consent.

Ages: 17 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2010-04; Primary Completion 2014-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Asthma Quality of Life Questionnaire with Standardized Activities [AQLQ(S)] | 12 months
  AQLQ(S) will be recorded at baseline, 6 months, and 12 months. The primary outcome will be the change in AQLQ(S) from baseline to 12 months.

SECONDARY OUTCOMES:
Asthma Control Questionnaire (ACQ) | 12 months
  The ACQ will be administered at baseline, 6 months, and 12 months. The secondary outcome will assess change in ACQ from baseline to 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Noseworthy, MD, Study Director — Alberta Children's Hospital; Rodel Padua, RRT, Study Director; Sheldon Spier, MD, Study Director — Alberta Children's Hospital; Ward Flemons, MD, Study Director — University of Calgary; Warren Davidson, MD, Principal Investigator — University of Calgary
Locations (1):
- Calgary Regional Pediatric Asthma Clinic, Calgary, Alberta, Canada